CLINICAL TRIAL: NCT01327833
Title: Cardiac Arrest Outcomes Data Evaluation
Brief Title: CODE Registry - Cardiac Arrest Outcomes Data Evaluation
Acronym: CODE
Status: Completed | Type: Observational
Sponsor: Instituto Dante Pazzanese de Cardiologia (Other)
Other Study IDs: IDPC-CODE
Record Dates: First submitted 2011-03-31; First posted 2011-04-04 (Estimated); Last update posted 2011-04-04 (Estimated); Status verified 2011-03

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Cardiac Arrest

SUMMARY:
The purpose of this study is based on method Utstein, registering all recommended items of that model, in addition to adding more information, characterizing this way using a template Utstein modified for the epidemiology of PCR-hospital in Brazil.

Objectives: establish a registry of patients suffering from respiratory (PCR)-hospital to assess demographic and clinical variables such as morbidity, mortality and standard practice in cardiopulmonary resuscitation (CPR). In addition, assess independent predictors associated with survival in several times and survival curves.

DETAILED DESCRIPTION:
Bedding: Despite of ongoing advances and standardizing worldwide trumpeted by CPR guidelines, yet is little knowledge of the effectiveness of procedures for intra and extra-hospital CPR, so vast are the opportunities for documentation of these results in the field of clinical and epidemiological research. Utstein style emerged, then as a proposed methodology for the PCR during the Conference held at the former monastery Utstein, Norway. The "Utstein Style" was also the model for the construction of the National Registry of Cardiac Pulmonary Resuscitation (NRCPR), sponsored by the American Heart Association (AHA). The proposal of this study is based on method Utstein, registering all recommended items of that model, in addition to adding more information, characterizing this way using a template Utstein modified for the epidemiology of PCR-hospital in Brazil.

Objectives: establish a registry of patients suffering from respiratory (PCR)-hospital to assess demographic and clinical variables such as morbidity, mortality and standard practice in cardiopulmonary resuscitation (CPR). In addition, assess independent predictors associated with survival in several times and survival curves.

Methods: Observational Study of prospective registration type, to document the clinical practice of cardiopulmonary resuscitation in-hospital effect in 17 hospitals and institutes of public and private Brazilian specialties. Additionally the longitudinal follow-up will be conducted until discharged, and measurement of mortality at 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Patient in cardiac arrest in-hospital
* Consent Form signed by subject's legally acceptable representative or by patient in case of survive

Exclusion Criteria:

* Patient in cardiac arrest out-hospital
* Cardiac arrest induced (e.g: for cardiac surgery)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients in cardiac arrest in-hospital in 17 hospitals and institutes of public and private Brazilian specialties.
Sampling Method: Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo, Brazil